CLINICAL TRIAL: NCT05167487
Title: Retrospective Observational Study of Resectable Stage IIIA Non-small Cell Lung Cancer Patients: Pathological Response After Neoadjuvant Treatment and Patient Outcomes
Brief Title: Pathological Response After Neoadjuvant Treatment on NSCLC
Acronym: PLANET
Status: Recruiting | Type: Observational
Sponsor: Fundación GECP (Other)
Responsible Party: Sponsor
Other Study IDs: GECP 21/03_PLANET
Record Dates: First submitted 2021-11-05; First posted 2021-12-22 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Stage IIIA Non-small Cell Lung Cancer
Keywords: Neoadjuvant Treatment; Observational study; Resectable IIIA patients; Non small cell lung cancer; Pathological response
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Carboplatin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: platinum-based neoadjuvant treatment and surgery.: Resectable stage IIIA non-small cell lung cancer patients treated with platinum-based neoadjuvant treatment and surgery.
  Interventions: Drug: Cisplatin; Drug: Carboplatin

INTERVENTIONS:
Drug: Cisplatin — Route of administration: Intravenous infusion. Neoadjuvant chemotherapy is often given 2 to 4 months before surgery.
  Other Names: Cis-diammine-dichloroplatinum; Platinol
Drug: Carboplatin — Route of administration: Intravenous infusion. Neoadjuvant chemotherapy is often given 2 to 4 months before surgery.
  Other Names: Paraplatin

SUMMARY:
This is a non-interventional, observational, multicenter and retrospective study. Being limited to the collection of patient data already filled in the Tumor Thoracic Registry data base and the data from stage IIIA clinical trials case report forms.

DETAILED DESCRIPTION:
This is a non-interventional, observational, multicenter and retrospective study that will not under any circumstances interfere in the physician's normal clinical practice. Being limited to the collection of patient data already filled in the Tumor Thoracic Registry (TTR) data base and the data from stage IIIA clinical trials case report forms, it does not entail any diagnostic or therapeutic procedure outside of normal clinical practice.

The primary objective is to assess pathological response after neoadjuvant treatment as a subrogate endpoint for overall survival and disease-free survival in resectable stage IIIA non-small cell lung cancer patients.

It is estimated that around 15-20 Spanish sites are enrolling patients with these characteristics in the TTR or in the stage IIIA clinical trials of the Fundación GECP.

Pathologists and physician's of these sites will be invited to participate in the PLANET study as all cases will be clinical-pathologically re-evaluated to reach the study objectives. Each pathologist will re-evaluate the specimens from the selected patients under common criteria.The sample size would be 150 patients enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with resectable stage IIIA disease (according to American Joint Committee on Cancer [AJCC] lung cancer edition 7 or 8) who were included in the Tumor Thoracic Registry data base and in stage IIIA clinical trials which the sponsor is Fundación GECP.
* Patients with histologically N2 involvement confirmed
* Patients diagnosed as stage IIIA from 2010 and 2017
* Patients who have received neoadjuvant platinum-based treatment and surgery
* Age ≥ 18 years at time of study entry
* PET /TC at diagnosis

Exclusion Criteria:

* Patients who received chemoradiotherapy neoadjuvant treatment
* Patients who were not resected after neoadjuvant treatment
* Patients who were diagnosed after June 2017

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include all resectable stage IIIA patients who have received platinum-based neoadjuvant treatment and surgery and that were diagnosed as stage IIIA from 2010 to 2017.The cohort of patients identified for the current study will be based on a portion of patients included in the Thoracic Tumor Registry (TTR) and in stage IIIA clinical trials approved by Spanish Health Authorities which the sponsor is Fundación GECP.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-12-13 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
To assess pathological response after neoadjuvant treatment as a subrogate endpoint for overall survival and disease-free survival in resectable stage IIIA non-small cell lung cancer patients. | From the end of neoadjuvant treatment until the last follow up or death, assessed up to 45 months
  Pathological response will be assessed as complete pathological response, major pathological response (defined as ≤10% of viable tumor cells) and incomplete pathological response.

SECONDARY OUTCOMES:
To describe the percentage of residual viable tumor in this population of patients under common criteria | From the end of neoadjuvant treatment until the last follow up or death,assessed up to 45 months
  A) No response or more than 70% of viable tumor: Lymph node major pathological response negative (LN-MPR)- B) ≤70% of viable tumor cells: Lymph node major pathological response positive (LN-MPR)+ C) No evidence of any viable tumor (including primary tumor): Complete pathological response
To describe the histopathological changes within tumor bed associated to tumor response | From the end of neoadjuvant treatment until the last follow up or death, assessed up to 45 months
  Types of histopathological changes within tumor bed: fibrosis, lymphoid aggregates and others
To correlate pathological response and post-surgical complications | From the end of neoadjuvant treatment until the last follow up or death, assessed up to 45 months
  Pathological response will be assessed as complete pathological response, major pathological response (defined as ≤10% of viable tumor cells) and incomplete pathological response.
To describe the relation between nodal downstaging after neoadjuvant treatment and overall survival | From the end of neoadjuvant treatment until the last follow up or death, assessed up to 45 months
  Downstaging after surgery is a reduction in the stage of a cancer. Overall Survival defined as the length of time from either the date of diagnosis or the start of the treatment that patients diagnosed with the disease are still alive.

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Provencio, MD, Study Chair — President of Grupo Español de Cáncer de Pulmón
Locations (17):
- Spain (17):
  - Hospital Universitario De A Coruna, A Coruña, A Coruña
  - Hospital General Universitario de Alicante, Alicante, Alicante
  - ICO Badalona, Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Vall d'Hebron, Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - ICO Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Insular de Gran canaria, Las Palmas de Gran Canaria, Gran Canaria
  - Hospital Dr. Negrín, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital 12 De Octubre, Madrid, Madrid
  - Hospital Universitario la Paz, Madrid, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitario Regional de Málaga, Málaga, Málaga
  - Complejo Hospitalario Universitario de Vigo, Vigo, Pontevedra
  - Hospital Universitario La Fe, Valencia, Valencia
  - Hospital Universitario Cruces, Barakaldo, Vizcaya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Web page of the sponsor where users can find more information about Fundación GECP studies — http://www.gecp.org